CLINICAL TRIAL: NCT06935695
Title: Surveillance Versus Prn bronChOscoPy aftEr aIrway stenTing (SCOPE-IT)
Brief Title: Surveillance Versus Bronchoscopy After Airway Stenting
Acronym: SCOPE-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Udit Chaddha, Associate Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY-24-01352
Record Dates: First submitted 2025-04-04; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Bronchial Stents
Keywords: Airway; Stent; Bronchoscopy; Surveillance
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surveillance Group (Experimental): Patients will be scheduled to undergo a surveillance bronchoscopy 4-6 weeks after the stent insertion.
  Interventions: Device: Bronchoscopy
- No Surveillance (Active Comparator): Patients will only undergo bronchoscopies if warranted by clinical symptoms deemed to be secondary to stent-related complications.
  Interventions: Device: Bronchoscopy

INTERVENTIONS:
Device: Bronchoscopy — Bronchoscopy is a procedure that uses a bronchoscope (a thin, tube-like instrument with a light and a lens for viewing) to examine the inside of the trachea, bronchi (air passages that lead to the lungs), and lungs. The bronchoscope is inserted through the nose or mouth.
  Other Names: PRN bronchoscopy

SUMMARY:
Randomized, pilot study that evaluates surveillance bronchoscopy versus no surveillance for patients that undergo tracheobronchial stenting

ELIGIBILITY:
Inclusion Criteria:

* All adult patients that undergo central airway (trachea, main stem bronchi and bronchus intermedius) stenting.

Exclusion Criteria:

* Inability to obtain informed consent due to cognitive, neurologic or psychiatric impairment.
* Lobar or segmental stents alone
* Terminally ill patients considered too sick to undergo a follow-up surveillance bronchoscopy
* Stent insertion as a trial for excessive central airway collapse (as the duration of these stents is only 1-2 weeks)
* Patients with a tracheostomy (as these patients can undergo frequent in-line suctioning that can affect the outcomes being assessed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of stent-related complications warranting an intervention | 3 months after enrollment
  Possible complications:
  Stent migration, biofilm formation, obstructive mucus plugging, obstructive granulation requiring intervention

SECONDARY OUTCOMES:
Number of unscheduled visits due to stent-related complications | 3 months after enrollment
  Number of unscheduled visits due to stent-related complications
Number of urgent care or emergency room visits due to stent-related complications | 3 months after enrollment
  Number of urgent care or emergency room visits due to stent-related complications
Number of hospitalizations due to stent-related complications | 3 months after enrollment
  Number of hospitalizations due to stent-related complications
Number of stent-related complications as detected during a bronchoscopy or on cross-sectional imaging | 3 months after enrollment
  Number of stent-related complications as detected during a bronchoscopy or on cross-sectional imaging
Protocol Feasibility Composite Score | 3 months after enrollment
  A composite score comprised from recruitment success (enrollment of target participant numbers), protocol adherence, data completeness, intervention safety, and resource availability to measure protocol feasibility. The total scale for the composite score is 1 to 5, with higher score indicating more feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Udit Chaddha, MBBS, Principal Investigator — Icahn School of Medicine
Locations (1):
- The Mount Sinai Health System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in Mount Sinai's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (to be determined).